CLINICAL TRIAL: NCT05783440
Title: Smartphone Reported Direct Patient Feedback on Postoperative Pain That is Directly Passed on to Surgical Ward Nurses, Effects on Patient Reported Postoperative Pain Outcomes and Pharmaco-therapy. A Prospective, Randomized, Single-blinded, Controlled Tria
Brief Title: Direct Patient Feedback on Postoperative Pain
Acronym: DPF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NL9697
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Applying a system in which patients undergoing surgery can report pain scores and other pain-related outcomes with their own smartphone, both during hospitalization and for three months after discharge. During clinical admission patient reported pain scores > 3 (NRS 0-10) in the intervention group are immediately passed on to the nurse who will receive a notification on a smartphone. In the control group the patients' pain scores are not sent to the nurse. After discharge, patients will report pain scores every two weeks for three months.
  Interventions: Behavioral: direct patient feedback
- control group (No Intervention): Participants in the control group report postoperative pain scores and other pain related outcomes with their own smartphone. Their reported pain-scores will not be surpassed to the nurses on the ward. All patient reported pain-scores by smartphone are stored in a database that is not accessible to medical or nursing staff from the nursing ward.

INTERVENTIONS:
Behavioral: direct patient feedback — Participants in the intervention group report postoperative pain scores and other pain related outcomes with their own smartphone. Pain scores reported by smartphone > 3 (NRS 0-10) are immediately passed on to the nurse who will receive a notification on a smartphone.
  All patient reported pain-scores by smartphone are stored in a database that is not accessible to medical or nursing staff from the nursing ward.
  Arms: Intervention group

SUMMARY:
Postoperative pain is common, can be severe, has a negative impact on outcomes after surgery and brings along major economic costs for society. A substantial part of patients may develop persistent post-surgical pain. Severity and duration of pain after surgery appear to have a role in this process but the transition from acute postoperative pain to chronic pain is only partially understood.

Effective treatment of postoperative pain is hampered by several barriers, including the way measurement of pain and registration of pain-scores are carried out by nurses in clinical practice. Modern technology offers new opportunities for pain measurement and direct patient feedback on postoperative pain, during and also after clinical admission. We developed a smartphone application that allows clinical patients to report pain scores and other pain related outcomes on postoperative pain with their own telephone device. Patient reported pain scores > 3 on a Numeric Rating Scale (NRS) 0-10 are immediately passed on to the nurse who receives a message of the reported pain score. This can lead to earlier detection of pain and a more timely treatment resulting in improved patient reported outcomes on postoperative pain

DETAILED DESCRIPTION:
Postoperative pain is common, can be severe, has a negative impact on outcomes after surgery and brings along major economic costs for society. A substantial part of patients may develop persistent post-surgical pain. Severity and duration of pain after surgery appear to have a role in this process but the transition from acute postoperative pain to chronic pain is only partially understood.

Effective treatment of postoperative pain is hampered by several barriers, including the way measurement of pain and registration of pain-scores are carried out by nurses in clinical practice. Modern technology offers new opportunities for pain measurement and direct patient feedback on postoperative pain, during and also after clinical admission. We developed a smartphone application that allows clinical patients to report pain scores and other pain related outcomes on postoperative pain with their own telephone device. Patient reported pain scores > 3 on a Numeric Rating Scale (NRS) 0-10 are immediately passed on to the nurse who receives a message of the reported pain score. This can lead to earlier detection of pain and a more timely treatment resulting in improved patient reported outcomes on postoperative pain

ELIGIBILITY:
Inclusion Criteria:

* Participants have to be 18 years or older
* Participants need to undergo a clinical surgical procedure for one of the three medical specialties mentioned above.
* Participants must be admitted to one of the participating surgical wards directly following discharge from the post anesthetic care unit after surgery.
* Participants have to stay admitted to the wards at least till the next day after surgery.
* Participants have to be in the possession of a smartphone that is able to receive a SMS text message and can sent data to a web based server.
* Participants must master the Dutch language and provide their written informed consent on forehand.
* Participants answered the first questionnaire (APS-POQ-R part I) before surgery.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Patients who do not wish to participate.
* Patients that for physical or cognitive impairments are unable to participate.
* Patients who do not possess a smartphone.
* Patients who are transferred to another ward during hospital admission e.g. the intensive care unit the first night after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient reported time in severe pain | every clinical admission day (8 a.m.-8 a.m.)
  Patient reported time in severe pain per separate clinical admission day (8 a.m.-8 a.m.), as reported by APS-POQ-R.

CONTACTS AND LOCATIONS:
Overall Officials: marjolein haveman, Study Chair — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No